CLINICAL TRIAL: NCT02342353
Title: A Phase I/II Study of Pacritinib in Patients With EGFR Mutant NSCLC After EGFR TKI
Brief Title: Pacritinib in Patients With Endothelial Growth Factor (EGFR) Mutant Non-small Cell Lung Cancer (NSCLC) After EGFR Tyrosine Kinase Inhibitor (TKI)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Drug shortage
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201503052
Record Dates: First submitted 2015-01-14; First posted 2015-01-19 (Estimated); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Non-Small Cell Lung Cancer; Nonsmall Cell Lung Cancer; Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase I (pacritinib and erlotinib) (Experimental): * Pacritinib will be administered orally twice a day; dosing will depend on the dose level the patient is enrolled.
  * Erlotinib will be taken by mouth on an outpatient basis daily at a dose of 150 mg.
  * A 28-day interval is defined as a cycle
  Interventions: Drug: Pacritinib; Drug: Erlotinib
- Phase II (pacritinib and erlotinib) (Experimental): * Pacritinib will be administered orally twice a day; the dose used will be the dose determined to be the MTD in phase I.
  * Erlotinib will be taken by mouth on an outpatient basis daily at a dose of 150 mg.
  * A 28-day interval is defined as a cycle
  Interventions: Drug: Pacritinib; Drug: Erlotinib

INTERVENTIONS:
Drug: Pacritinib
  Other Names: SB1518
Drug: Erlotinib
  Other Names: Tarceva®; OSI-774

SUMMARY:
The goal of the study is to find the best dose of pacritinib when given in combination with erlotinib.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic or unresectable locally advanced NSCLC with known sensitive EGFR mutations. Patients with mutations in T790M are eligible if they have progressed after treatment with a third generation EGFR tyrosine kinase inhibitor (osimertinib), but otherwise patients must have EGFR T790M negative or unknown status. Patients previously treated with third generation EGFR tyrosine kinase inhibitor must have achieved a treatment benefit of at least 4 months.
* Disease progression following therapy with erlotinib, afatinib, or gefitinib
* May have received one or more prior treatments with chemotherapy
* Measurable disease defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 10 mm with CT scan, as ≥ 20 mm by chest x-ray, or ≥ 10 mm with calipers by clinical exam.
* At least 18 years of age.
* ECOG performance status ≤ 1
* Normal bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1,500/mcl
  * Platelets ≥ 100,000/mcl
  * Hemoglobin ≥ 9.0 g/dL
  * Total bilirubin ≤ 2.0 x IULN
  * AST (SGOT) / ALT (SGPT) ≤ 3.0 x IULN; if liver metastases, ≤ 5.0 x IULN
  * Serum creatinine ≤ 1.5 x ULN
* Adequate cardiac function as demonstrated by LVEF ≥ 50% performed no more than 4 weeks prior to enrollment.
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Able to swallow pills
* Able to understand and willing to sign a Human Research Protection Office (HRPO) approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Known pre-existing interstitial lung disease.
* Leptomeningeal carcinomatosis or other untreated or symptomatic central nervous system (CNS) metastases. Patients with asymptomatic CNS metastases, other than leptomeningeal disease, are eligible provided they have been clinically stable without requiring increase in steroid dose for at least 4 weeks.
* A history of other malignancy ≤ 5 years previous with the exception of basal cell or squamous cell carcinoma of the skin which were treated with local resection only or carcinoma in situ of the cervix.
* Received any chemotherapeutic or targeted agent (approved or investigational) for NSCLC within 2 weeks of initiation of pacritinib (with the exception of erlotinib).
* Currently receiving any other investigational agents.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to pacritinib or other agents used in the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and/or breastfeeding: Patient must have a negative pregnancy test within 14 days of study entry.
* Known HIV-positivity on combination antiretroviral therapy because of the potential for pharmacokinetic interactions with pacritinib. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
* Use of potent cytochrome P450 3A4 (CYP3A4) inducer within one week of pacritinib initiation
* Patients with CTCAE grade 2 cardiac arrhythmias may be considered for inclusion if the arrhythmias are stable, asymptomatic, and unlikely to affect patient safety. Patients will be excluded if they have ongoing cardiac dysrhythmias of CTCAE grade ≥ 3, corrected QT interval (QTc) prolongation >450ms, or other factors that increase the risk for QT interval prolongation (eg, heart failure, hypokalemia [defined as serum potassium <3.0mEq/L that is persistent and refractory to correction], or family history of long QT interval syndrome).
* Any gastrointestinal (GI) or metabolic condition that could interfere with absorption of oral medication such as ongoing grade 3 or higher diarrhea, constipation, nausea, or vomiting.
* Active viral hepatitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-05-18 (Actual); Primary Completion 2018-02-06 (Actual); Study Completion 2018-02-06 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicities and maximum tolerated dose (MTD) - Phase I only | Completion of cycle 1 of all Phase I patients (estimated to be 1 year)
  The maximum tolerated dose (MTD) is defined as the dose level immediately below the dose level at which 2 patients of a cohort (of 2 to 6 patients) experience dose-limiting toxicity during the first cycle. Dose escalations will proceed until the MTD has been reached.
  A patient is evaluable for DLT assessment only during Cycle 1 of treatment. If the patient is not able to be treated on Day 1 of Cycle 2, then s/he is still considered in Cycle 1 active treatment and can experience a DLT. Once the patient has been treated in Cycle 2, s/he will no longer be evaluated for DLTs in all subsequent cycles.
Response rate - Phase II only | Up to 5 years
  * Partial response + complete response per RECIST 1.1 criteria
  * Study terminated prior to enrolling any phase II participants
  * Complete response (CR) = disappearance of all target lesions, non-target lesions, and normalization of tumor marker level
  * Partial response (PR) = at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline of sum diameters

SECONDARY OUTCOMES:
Adverse events (toxicities) | 30 days post completion of treatment (estimated to be 9 months)
  The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for all toxicity reporting.
Disease control rate (DCR) | Up to 5 years
  Percentage of patients who achieve complete response, partial response, or stable disease per RECIST 1.1 criteria.
  * Complete response (CR) = disappearance of all target lesions, non-target lesions, and normalization of tumor marker level
  * Partial response (PR) = at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline of sum diameters
  * Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Progression-free survival (PFS) | Up to 5 years
  * PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
  * Progressive disease (PD) = at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study, appearance of one or more non-target lesion(s) and/or unequivocal progression of existing non-target lesions
Overall survival (OS) | Up to 5 years
  Overall survival is defined as the time interval from date of diagnosis to date of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Morgensztern, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu